CLINICAL TRIAL: NCT03538964
Title: Assessing the Astigmatism Reducing Effect With Toric IOLs in Eyeswith Low Astigmatism
Acronym: Low Asti
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Low Asti
Record Dates: First submitted 2018-04-30; First posted 2018-05-29 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Cataract; Astigmatism
Keywords: Cataract; Low Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toric intraocular lens (IOL) (Active Comparator): toric intraocular lens for low astigmatism correction
  Interventions: Procedure: toric intraocular lens
- Non toric intraocular lens (IOL) (Sham Comparator): non toric intraocular lens
  Interventions: Procedure: non toric intraocular lens

INTERVENTIONS:
Procedure: toric intraocular lens — cataract surgery with implantation of an toric intraocular lens
  Arms: Toric intraocular lens (IOL)
Procedure: non toric intraocular lens — cataract surgery with implantation of a non toric intraocular lens
  Arms: Non toric intraocular lens (IOL)

SUMMARY:
Comparison of the astigmatism reducing effect of a toric IOL with a non toric IOL in eyes with low corneal astigmatism.

DETAILED DESCRIPTION:
With increasing demands of patients concerning refractive outcome after cataract surgery, toric intraocular lenses (IOLs) that correct corneal astigmatism have been introduced more widely to cataract surgery. Originally, toric IOLs were used mainly for patients with high degrees of astigmatism. Since a couple of years, toric IOLs are available from numerous manufacturers to correct moderate amounts of astigmatism which are much more prevalent with about 8% having a corneal astigmatism of 2.0D or more in the cataract population. 5Using toric IOLs for these eyes results in less spectacle dependence of patients due to the astigmatic correction. Other astigmatism reducing techniques, such as peripheral corneal relaxing incisions and opposite clear corneal incisions were shown to be less predictable. Although the use of toric IOLs became the gold standard to correct corneal astigmatism during cataract surgery , there is still uncertainty, if low astigmatism should be corrected. Visser et al. showed that moderate astigmatism of than 1.5D should be corrected for monofocal IOLs and Hayashi showed that remaining astigmatism of 1.0D already decreases visual quality in eyes with multifocal IOLs. Although correction of low corneal astigmatism appears to be beneficial, some hurdles have to be taken into account. In eyes with low corneal astigmatism the accuracy of measuring the astigmatism meridian is relatively low. Furthermore, different corneal measurement techniques are not always comparable and it is difficult to know, which device shows the correct amount of astigmatism. Additionally, the correction of the spherical equivalent is of high importance, as a refractive surprise will also attenuate the astigmatism reducing effect of the toric IOL. Aim of this study is to assess, if toric IOLs are useful in patients with low amounts of corneal astigmatism and to quantify the sources of error in toric IOL power calculation.

ELIGIBILITY:
Inclusion Criteria:

* cataract
* Age 21 and older
* Regular corneal astigmatism 0.5D up to 1.5 D and difference between eyes not more than 0.75D
* written informed consent prior to surgery

Exclusion Criteria:

* relevant other ophthalmic diseases such as: pseudoexfoliation, glaucoma, traumatic cataract corneal scars, and other co-morbidity that could affect capsule bag stability ( e.g. Marfan syndrome)
* Irregular corneal astigmatism on corneal topography
* In case of pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2020-05-02 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Subjective refraction to detect remaining astigmatism (in Diopters) between both groups | 12 months

SECONDARY OUTCOMES:
Biometrical measurement of axial length (in mm), anterior chamber depth (in mm), corneal astigmatism (radii and axial degrees) | 12 months
Purkinjemeter measurement of Tilt (in degrees) and Decentration (in degrees) of the intraocular lens | 12 months
Wavefront analysis of high order aberrations (root mean square, in microns) | 12 months
Questionnaire to asses patients subjective satisfaction with visual outcome | 12 months
  In the questionnaire the patient has to choose if different tasks (e.g. reading, driving, watching TV) are easier for him/ her with the right eye, the left eye, or if there is no difference between both eyes

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided